CLINICAL TRIAL: NCT02868619
Title: Binge Eating Disorder and Obesity : Reward System Abnormalities in Response to Food Stimuli and Research Operability by Deep Brain Stimulation Criteria: Functional MRI Study
Brief Title: Binge Eating Disorder and Obesity : Functional MRI Study
Acronym: BED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9093
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Binge Eating Disorder; Obesity
Keywords: fMRI; Deep brain stimulation; Food; Eating; Reward
MeSH Terms: conditions — Binge-Eating Disorder; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy controls (Other): Non obese adolescents without Binge Eating Disorder (BED)
  Interventions: Other: Functional MRI; Other: ADO-BEDS scale; Other: R-CMAS scale
- Patients with BED (Other): Obese adolescents with BED with Binge Eating Disorder (BED)
  Interventions: Other: Functional MRI; Other: ADO-BEDS scale; Other: R-CMAS scale

INTERVENTIONS:
Other: Functional MRI — functional MRI assessed on all the volunteers in condition of hunger and in Condition of satiety
Other: ADO-BEDS scale — Evaluate the severity of BED according to Marcus and Kalarchian temporary diagnosis criteria
Other: R-CMAS scale — Evaluate the anxiety

SUMMARY:
Obesity, defined as BMI> 30kg / m2, is a major public health problem, with devastating medical and psychological consequences. 30% of obese suffer from BED type of eating disorders. The optimal treatment of obesity remains bariatric surgery, failed in 20% of cases. Many arguments are in favor of the involvement of the reward circuitry, with the central role of NAc in the pathophysiology of BED and obesity. The recent application and effectiveness of DBS (Deep Brain Stimulation) in refractory psychiatric disorders suggest that DBS may be of interest in treating obesity and BED with potential target for the NAc. This project propose to study fMRI activation of the reward system in response to food stimuli to better direct the DBS targets. This is a pilot study to define indication criteria based on fMRI to obese BED patients are potential candidates for treatment with DBS.

DETAILED DESCRIPTION:
The aim of this functional neuroimaging study is to analyze brain responses to visual food cues in obese (body mass index > 97th percentile) adolescents with BED (according to the criteria Marcus and Kalarchian) compared with healthy control adolescents in two situations : hunger et satiety.

Fifteen obese adolescents (12/16 years) with BED and fifteen healthy control adolescents will be enrolled in the study protocol. Participants will be instructed not to eat food for at least 6 hours prior to the first imaging session. After the initial set of functional and anatomic scans, participants will be fed a standard calorie meal. Approximately 1 hour later, the experiment will be repeated while participants are in a satiated condition. The cortical fMRI activation will be measured during the following four experimental visual conditions : high calory food, low calory food, disgust and neutral presented in block design.

First-level and second-level differences in neural activation assessed during functional MRI in the different conditions will then be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Non specific inclusion criteria

  * Age limits ≥ 12 et < 16 years
  * Collection of the informed consent. For the minor patients, signature of parents
  * Affiliation or recipient with the mode of social security.
  * No associated evolutionary pathologies
* Specific inclusion criteria for the patients

  * Existence of a current food disorder of the conducts of type binge eating disorder according to the criteria Marcus and Kalarchian
  * Diagnosis of obesity defined by a body mass index > 97th percentile
  * Severity criteria defined by: Evolution of the obesity and the BED for at least 5 years AND Not answer to a dietary, pharmacological, psychotherapeutic care during at least 6 months
* Specific inclusion criteria for the volunteers

  * Absence of a current food disorder of the conducts of type binge eating disorder according to the criteria Marcus and Kalarchian
  * Absence of antecedent of neurological disorder
  * an actual body mass index < 90th percentile

Exclusion Criteria:

* IRM contraindication
* Pacemaker
* Port(Bearing) of surgical clips in the cervico-cephalic region or implanted medical surgical material(equipment) susceptible to mobilize under the influence of magnetic gradients
* Intraocular foreign body
* Metalic foreign body
* claustrophobia
* The existence of possible psychiatric histories will be individually estimated
* Pregnancy and breastfeeding
* Loss of liberty by court or administrative order

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2014-12-05 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Differences in neural activation assessed during functional MRI | 4 years
  The main objective of this study is the identification in patients with obesity and Binge Eating Disorder (BED) of functional MRI activation profiles (reward system) in response to food stimuli. The activation profiles will be analyzed by varying physiological conditions of hunger and satiety, and motivational value attributed to the food (calorie).

SECONDARY OUTCOMES:
Pairwise comparisons in neural activation assessed during functional MRI | 4 years
  Further pairwise comparisons in neural activation assessed during functional MRI help to define DBS indication criteria / operability for BED obese candidates.

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne CYPRIEN, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Chu Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charroud C, Poulen G, Sanrey E, Menjot de Champfleur N, Deverdun J, Coubes P, Le Bars E. Task- and Rest-based Functional Brain Connectivity in Food-related Reward Processes among Healthy Adolescents. Neuroscience. 2021 Mar 1;457:196-205. doi: 10.1016/j.neuroscience.2021.01.016. Epub 2021 Jan 21. PMID 33484819
- [Derived] Charroud C, Menjot de Champfleur N, Sanrey E, Pfeuffer J, Deverdun J, Le Bars E, Coubes P. Differential effects of hunger on cerebral blood flow in healthy adolescents. Behav Brain Res. 2020 Apr 6;383:112505. doi: 10.1016/j.bbr.2020.112505. Epub 2020 Jan 23. PMID 31982461